CLINICAL TRIAL: NCT00264394
Title: Efficacy of a Computerised Physician Reminder System to Control Cardiovascular Risk Factors in HIV-infected Patients Receiving Antiretroviral Therapy: A Nested Randomised Controlled Cluster Trial Within the Swiss HIV Cohort Study
Brief Title: Cardiovascular Risk Factor Management in HIV Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SNF 3345-062041 SHCS 480; 480 (Other: Swiss HIV Cohort Study Registry); 480 (Other: Swiss HIV Cohort Study)
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Heart Disease; Dyslipidemia; Diabetes Mellitus, Non-Insulin-Dependent; HIV Infection
Keywords: Computer generated reminder system; quality control; dyslipidemia; antiretroviral therapy; HIV infection
MeSH Terms: conditions — Coronary Disease; Dyslipidemias; Diabetes Mellitus, Type 2; HIV Infections | interventions — Guidelines as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Updated CHD risk profiles (Experimental): Provision of regularly updated CHD risk profiles
  Interventions: Behavioral: Updated CHD risk profiles
- Guidelines (Active Comparator): Physicians received guidelines only
  Interventions: Behavioral: Guidelines

INTERVENTIONS:
Behavioral: Updated CHD risk profiles — Provision of computer generated CHD risk profiles
  Other Names: Computer assisted intervention to reduce CHD risk
  Arms: Updated CHD risk profiles
Behavioral: Guidelines — provision of guidelines for CHD risk factor management only
  Other Names: guidelines group
  Arms: Guidelines

SUMMARY:
There is growing evidence that antiretroviral therapy (ART) increases the risk of coronary heart disease (CHD) through metabolic side effects, such as dyslipidemia, insulin resistance, and type II diabetes. Prevalence of risk factors for CHD in HIV-infected individuals receiving ART in the Swiss HIV Cohort Study (SHCS) is high. This cluster randomised controlled trial is nested into the SHCS and will investigate whether physicians randomised to the routine provision of risk profiles from their patients receiving ART will improve the management of risk factors in HIV-infected patients compared to control physicians not routinely receiving such information. Risk profiles will be generated by the SHCS data center and provided to clinicians in all study centers.

DETAILED DESCRIPTION:
Evidence from the D.A.D. study, an international cohort study which includes a large proportion of SHCS patients, suggests that exposure to antiretroviral therapy (ART) increases the risk of coronary heart disease (CHD) most likely due to ART induced metabolic changes like dyslipidemia, insulin resistance, and type II diabetes. The exact mechanisms for these metabolic changes and whether specific classes or combinations of ART are causally related to these changes are not known. Of males aged < 40 and > 40 years in the SHCS, 8.8% and 32.5% are at moderate (10% - 20%) and 1.7% and 6.9% at high (≥ 20%) risk of CHD in 10 years according to the Framingham algorithm. The overall percentage at moderate and high 10-year risk of CHD was 14.9% and 3.0%, respectively. Therefore, an intervention to reduce CHD risk among individuals at high risk for CHD is warranted. We propose a randomised controlled cluster intervention trial to reduce total cholesterol in all HIV-infected individuals in the SHCS (primary endpoint) and in those with greater than or equal to 10% 10 year risk of CHD based on the Framingham score (secondary endpoint). The intervention is the receipt of structured continuously updated information on CHD risk factors and treatment of CHD risk factors of HIV-infected patients. Randomisation will be done at the physician level and stratified by centre (7 centres of the SHCS, outpatient clinic or hospital), and size of patient volume for registered private practices. For physicians randomised to the intervention group, a flow sheet with information on risk factors and treatment status of CHD will be provided for each of their patients every 6 months by the SHCS data centre. Each centre and each physician treating SHCS patients will receive internationally and locally approved guidelines for the management of risk factors for CHD in HIV-infected patients. The intervention will be limited to 18 months. Our goal is a 7% reduction in total cholesterol (primary endpoint) between the intervention and the control group in the entire cohort. With alfa-error of 5%, power of 80% and a loss to follow-up of 10%, 408 patients per arm will be needed. Sample size calculations adapted to the cluster design of the trial show that we have sufficient power to detect a 12% reduction in total cholesterol in patients receiving ART and at moderate to high risk of CHD. Further secondary endpoints are a reduction of systolic and diastolic blood pressure and of overall Framingham risk score. We will additionally monitor whether changes in ART due to high risk of CHD, or treatment of CHD risk factors decreases the proportion of patients with non-sustained control of HIV-viremia. Data from this nested cluster trial will provide important information as to whether provision of an individual's CHD profile will improve monitoring and reduce CHD risk factors in HIV-infected patients in the SHCS.

ELIGIBILITY:
Inclusion Criteria:

For analysis of the primary endpoint:

* All individuals in the SHCS

  * aged 18 or older
  * have a cohort visit in the 12 months preceding the randomisation date with a complete baseline dataset on CHD risk factors

For analysis of secondary endpoints:

* All individuals in the SHCS

  * aged 18 or older
  * have a cohort visit in the 12 months preceding the randomisation date with a complete baseline dataset on CHD risk factors
  * at least 3 months of ART and at moderate to high risk of CHD (10% 10 years risk of CHD according to the Framingham risk score).

Exclusion Criteria:

* Pregnant females
* Patients in the SHCS not receiving ART

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4097 (Actual)
Dates: Start 2006-07; Primary Completion 2008-10 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Reduction in total cholesterol in the entire SHCS population | 18 months

SECONDARY OUTCOMES:
The reduction in total cholesterol, systolic and diastolic blood pressure, and Framingham 10-year CHD risk score in individuals with a greater than or equal to 10% 10 year risk of CHD (according to the Framingham risk profile) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Heiner C Bucher, MD, Principal Investigator — Basel Institute for Clinical Epidemiology University Hospital Basel
Locations (7):
- Switzerland (7):
  - University Hospital Basel, Basel, Canton of Basel-City
  - Division des Maladies Infectieuses, Hopital Universitaire Geneve, Geneva, Canton of Geneva
  - Division Maladies Infectieuses, Hopital Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud
  - Departement Innere Medizin Kantonsspital St. Gallen, Sankt Gallen, Canton Saint Gall
  - Ospedale Civico Lugano, Lugano, Canton Ticino
  - Abteilung für Infektionskrankheiten & Spitalhygiene, Universitätsspital Zürich, Zurich, Canton Zurich
  - Klinik und Poliklinik für Infektiologie, Inselspital, Bern

REFERENCES:
- [Background] Bucher HC, Rickenbach M, Young J, Glass TR, Vallet Y, Bernasconi E, Cavassini M, Fux C, Schiffer V, Vernazza P, Weber R, Battegay M; Swiss HIV Cohort Study. Randomized trial of a computerized coronary heart disease risk assessment tool in HIV-infected patients receiving combination antiretroviral therapy. Antivir Ther. 2010;15(1):31-40. doi: 10.3851/IMP1475. PMID 20167989
- See also: Swiss HIV Cohort Study — http://www.shcs.ch